CLINICAL TRIAL: NCT06396728
Title: Use of GI BIOTICS 100B UFC to Improve Intestinal Health and Sports Performance in Older Adults
Brief Title: Use of GI BIOTICS 100B UFC to Improve Intestinal Health in Older Adults
Acronym: GIBIOTICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Borja Martínez Tellez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: TRFE-SI-2023/006
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Gut Microbiota; Gut Health; Digestive System; Intestinal Inflammation; Strength
Keywords: Gut; Health; Digestive System; Intestinal Inflammation; Strength

STUDY DESIGN:
Intervention Model Description: The study involves a total of 44 men who will be randomly selected to be part of two groups: one who will consume a placebo capsule and another who will consume GI BIOTICS 100B UFC daily for a period of 8 weeks.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consumption of GI BIOTICS 100B UFC (Experimental): Participants will consume one GI BIOTICS 100B UFC capsule daily for a period of 8 weeks; n=22.
  Interventions: Dietary Supplement: GI BIOTICS 100B UFC
- Placebo Consumption (Placebo Comparator): Participants will consume one placebo capsule daily for a period of 8 weeks; n=22.
  Interventions: Dietary Supplement: Placebo Consumption

INTERVENTIONS:
Dietary Supplement: GI BIOTICS 100B UFC — Consumption of GI BIOTICS 100B UFC.
  Arms: Consumption of GI BIOTICS 100B UFC
Dietary Supplement: Placebo Consumption — Consumption of a placebo capsule.
  Arms: Placebo Consumption

SUMMARY:
Type of study: Clinical Trial.

Main objective: To study the effect of daily consumption of the probiotic (GI BIOTICS 100B UFC) on intestinal inflammatory markers, intestinal microbiota, intestinal health, body composition and sports performance in older adults for 8 weeks.

Participant Population/Health Conditions: The study will involve 44 sedentary men with a body mass index > 25 kg/m2 and aged between 60 and 75 years.

Participants Will:

Be randomised into one of two groups: consumption of a placebo capsule (comparison group) and consumption of GI BIOTICS 100B UFC daily for a period of 8 weeks (experimental group). Provide feces and blood samples before and after the 8-week intervention. Undergo analysis of these samples using advanced techniques to understand the effect of the consumption of the probiotic. Undergo a submaximal stress test and muscle strength will be measured using a handgrip dynamometer.

DETAILED DESCRIPTION:
Intestinal health is essential for the general well-being of the body given the great diversity of microorganisms known as intestinal microbiota that the intestine houses. These microorganisms play a crucial role in digestion, nutrient absorption, metabolism and regulation of the immune system. However, various factors such as an unbalanced diet, stress and the use of antibiotics or other medications can alter the balance of the microbiota and lead to intestinal health problems, as occurs in those over 60 years of age. In this context, the use of probiotics has gained recognition as an effective strategy to improve intestinal health. Probiotics involve inoculating the intestine with live microorganisms that, when consumed in adequate amounts, provide health benefits. These beneficial bacteria for our body can colonize the intestine, restore the balance of the microbiota and promote an environment conducive to the proper functioning of the digestive system. Probiotics have shown evidence of improving gut health by strengthening the intestinal barrier, reducing intestinal permeability, and decreasing inflammation. In addition, they can improve the digestion of certain foods, produce beneficial vitamins and metabolites, and compete with harmful bacteria to occupy space in the intestine. Recently, it has been shown that specific bacterial species in the intestine could improve exercise capacity in athletes. In this line of thinking, novel and unpublished data from our laboratory unequivocally demonstrate that specific bacterial species can improve exercise capacity in mice through the gut-muscle axis as the main underlying mechanism. That being said, we hypothesize that daily consumption of the probiotic GI BIOTICS 100B UFC, designed by HSN, will reduce intestinal inflammation by improving gut microbiota composition and gut health. Furthermore, this improvement in the intestinal microbiota will reduce the percentage of body fat, improving the ability to run to exhaustion and force generation in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 60-75 years of age men. BMI >25 kg/m2. Be willing to be randomized to either of these 2 groups. Must be sedentary (i.e., do not exercise or go to the gym).
* Must be willing to adhere to all study procedures, including attendance at all study visits.
* Must be willing to have biological samples stored for future research.
* Having self-defined digestive problems (poor digestions, constipation, bloating in response to food, refluxes, heartburn)

Exclusion Criteria:

* Diabetes Mellitus
* High Blood Pressure
* Being intolerant to lactose, fructose or sorbitol
* Having consumed probiotics or antibiotics in the last 3 weeks
* Be a regular smoker

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Intestinal permeability | 1 year
  LPS and Zonulin will be quantified in feces before and after the intervention
Gut microbiota | 1 year
  In feces samples, 16S ribosomal RNA sequencing will be performed to quantify the composition of the intestinal microbiota.

SECONDARY OUTCOMES:
Body composition | 1 year
  The body composition of the participants will be measured using a state-of-the-art device.
Blood samples | 1 year
  These samples will be centrifuged, and the serum and plasma will be aliquoted and stored at -80ºC for future analyses.
Submaximal physical effort test | 1 year
  Sports performance will be evaluated through a submaximal physical effort test.
Muscle strength | 1 year
  Muscle strength will be measured using a handgrip dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain